CLINICAL TRIAL: NCT00815685
Title: A Pilot Study of Eicosapentaenoic Acid (EPA) in Patients With Cancer Cachexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15190
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Results first posted 2011-09-08 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2013-12

CONDITIONS: Cancer Cachexia
Keywords: n-3 fatty acids; nutritional treatment; molecular pathogenesis
MeSH Terms: interventions — Eicosapentaenoic Acid; Omacor; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eicosapentaenoic Acid (Experimental)
  Interventions: Drug: Eicosapentaenoic Acid

INTERVENTIONS:
Drug: Eicosapentaenoic Acid — Participants will receive Lovaza at a dose of 4 g for 6 weeks. Participants will be examined at six weeks for change in protein status as indicated by change in morphological (Height, weight, body mass index, body composition, lean body mass, body fat %), and biochemical (serum prealbumin) markers of protein status and immunological cytokines (Il-6, TNF- α) markers implicated in cancer cachexia. At baseline, 3 and 6 weeks, participants will undergo interviews and laboratory analysis for determining compliance and treatment-related toxicity.
  Other Names: Lovaza; EPA; omega-3-acid ethyl esters; docosahexaenoic acid; DHA

SUMMARY:
The data collected through this pilot study will allow us to increase our understanding of cancer cachexia and the effect of Eicosapentaenoic Acid (EPA) on cancer cachexia. Our long-term goal is to improve nutritional treatment and reduce illness in the cancer patient population.

DETAILED DESCRIPTION:
People who have cancer can get what is called cancer cachexia (CC). The symptoms of CC include getting full quickly when eating (early satiety), loss of appetite, weakness resulting in weight loss and loss of lean body mass. Even a weight loss of 5% in cancer patients reflects poor health, hospitalization, and a higher rate of illness. Research shows that the elderly are at higher risk for deficiency of vitamins and trace minerals. Other pre-existing chronic diseases and drug therapies in this population may increase the needs of certain nutrients. Recent studies have also shown that advanced malnutrition is much more difficult to treat in the elderly than in younger adults, and the consequences of failure to treat it delays recovery and can decrease function and quality of life. At this time, the ways to treat CC include giving medications to increase appetite and giving nutritional supplements that are high in calories and protein.

Recent studies have shown that certain types of fats that are present in fish, walnuts and other foods that we eat called Eicosapentaenoic acid (EPA) may help with weight gain, especially gain in muscle and improve quality of life in patients with pancreatic cancer. However, EPA has never been studied in prevention of cancer cachexia in cancer patients showing early signs of weight loss. Based on these early, small studies, it is clear that we need to study if and how EPA can prevent loss of muscle and weight in cancer patients and prevent this from becoming worse.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women 25-80 years of age (inclusive)
* Confirmed diagnosis of Cancer (other than pancreatic cancer) Unintentional weight loss of >5% of body weight within 3 months of admission to the study
* Use of effective means of contraception (men and women) in patients of child-bearing potential
* Normal baseline liver function tests (LFTs) as determined by alanine aminotransferase (ALT) levels. Common Toxicity Criteria (CTC)) version 3 grade 1 elevation in ALT (>Upper Limit of Normal[UNL]-2.5 x UNL) withhold admitting participant to the study until recovery to normal; LFTs will be considered valid for consideration of eligibility if drawn within the previous 2 weeks, otherwise new labs will be drawn.
* Able and willing to give written informed consent : Each participant must be aware of the nature of his current medical condition and must be willing to give consent after being informed of the experimental nature of therapy, alternatives, potential benefits, side-effects, risks and discomforts.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0- 2 (Karnofsky score >60%)
* Concurrent use of coumadin or warfarin is okay. The follow-up monitoring for prothrombin (PT), partial thromboplastin time (PTT) and International Normalized Ratio (INR) for patients on warfarin and/or coumadin will follow the standard of care as dictated by the prescribing physician. If the prescribing physician is not a Moffitt physician, then the prescribing physician will be notified by the research staff of the subject participating in the study, and monitors for PT, PTT and INR will be obtained from patient during the 6 week study for review.

Exclusion Criteria:

* Patients with current diagnosis or history of pancreatic cancer
* Current use of anticoagulants other than coumadin, warfarin, or aspirin
* Use of other nutritional supplements other than multivitamins and minerals
* Allergy to fish or seafood
* Using Marinol or Megace
* Known history of hepatic or renal disease
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation or study drug administration, or may interfere with interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Evidence of bleeding diathesis or coagulopathy
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation or study drug administration, or may interfere with interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study
* Pregnant (positive pregnancy test) or lactating

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Kumar, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - Martin Memorial, Stuart, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants will include cancer patients with Men and Women >25 years of age (inclusive), with a confirmed diagnosis of cancer, unintentional weight loss of >5% of body weight, using uniform established diagnostic criteria and be admitted to the study within 3 month of diagnosis.
Groups:
- Eicosapentaenoic Acid (Lovaza): Participants to receive Lovaza at a dose of 4 g for 6 weeks.
Period: Overall Study
Arm/Group | Eicosapentaenoic Acid (Lovaza)
Started | 36
Completed | 14 (Complete pre and post-treatment serum samples were available for 14 participants.)
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Eicosapentaenoic Acid (Lovaza)
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Albumin
Description: Change in protein status at 6 weeks after initial diagnosis of weight loss of >5% body weight as indicated by morphological, biochemical and immunological intermediate biomarkers.
Time Frame: 6 weeks per patient
Measure: Median (Full Range); unit: g/dL
Arm/Group | Eicosapentaenoic Acid (Lovaza)
Number analyzed (Participants) | 14
g/dL | 4.0 [3.10 to 4.70]

2. Secondary Outcome: Number of Participants With Proteasome Activity That Was Inhibited in the Range of 6%-29%.
Description: There is no expected range for "normal" activity since there is not currently a clinical indication for these molecular markers. Comparison of ranges can be made between groups (such as those that received treatment and not). This was an exploration of potential in the pilot study and further research is indicated to better understand the metabolic abnormalities observed in cancer cachexia as well as potential benefits of using agents such as EPA.
Time Frame: 6 weeks per patient
Population: Participants with available pre and post-treatment serum samples.
Measure: Number; unit: Participants
Arm/Group | Eicosapentaenoic Acid (Lovaza)
Number analyzed (Participants) | 14
Participants | 9

ADVERSE EVENTS:
Time Frame: 6 weeks per participant
Arm/Group | Eicosapentaenoic Acid (Lovaza)
Serious Adverse Events (participants affected / at risk) | 4/36
Other Adverse Events (participants affected / at risk) | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eicosapentaenoic Acid (Lovaza) (N=36)
CNS (Vascular disorders) | 1 (1) — Grade 3 - unrelated
Dehydration (Gastrointestinal disorders) | 2 (2) — Grade 3 - unrelated
Diarrhea (Gastrointestinal disorders) | 2 (2) — Grade 3 - unrelated
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3 - unrelated
Febrile Neutropenia (General disorders) | 2 (2) — Grade 3 - unrelated
Glucose serum-high (Metabolism and nutrition disorders) | 1 (1) — Grade 3 - unrelated
Hypotension (Cardiac disorders) | 1 (1) — Grade 3 - unrelated
Mucositis/stomach - Oral cavity (Gastrointestinal disorders) | 1 (1) — Grade 3 - unrelated
Nausea (Gastrointestinal disorders) | 2 (2) — Grade 3 - unrelated
Pain - Chest/Thorax (General disorders) | 1 (1) — Grade 3 - unrelated
Pain - abdomen (General disorders) | 1 (1) — Grade 3 - unrelated
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3 - unrelated
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3 - unrelated
Potassium serum-low (Metabolism and nutrition disorders) | 2 (2) — Grade 3 - unrelated
Vomitting (Gastrointestinal disorders) | 2 (2) — Grade 3 - unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eicosapentaenoic Acid (Lovaza) (N=36)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) — Grade 1-3 - unrelated
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2) — Grade 1 - unlikely to be related
Anorexia (Gastrointestinal disorders) | 5 (6) — Grade 1-3 - unlikely to be related
Bruising in absence of Grade 3 or 4 thrombocytopenia (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1 - unlikely to be related
Constipation (Gastrointestinal disorders) | 2 (2) — Grade 1-3 - possibly related
Constipation (Gastrointestinal disorders) | 1 (1) — Grade 2 - unlikely to be related
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 2 - possibly related
Diarrhea (Gastrointestinal disorders) | 2 (3) — Grade 1 - unlikely to be related
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) — Grade 1 - unlikely to be related
Dizziness (General disorders) | 2 (2) — Grade 1-3 - unlikely to be related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Grade 1-3 - unlikely to be related
Edema: limb (Blood and lymphatic system disorders) | 1 (1) — Grade 2 - unrelated
Fatigue (General disorders) | 11 (13) — Grade 1-3 - unlikely to be related
Glucose, serum-high (Metabolism and nutrition disorders) | 1 (1) — Grade 1-3 - unrelated
Hair loss (Skin and subcutaneous tissue disorders) | 5 (6) — Grade 1-3 - unlikely to be related
Hemoglobin (Blood and lymphatic system disorders) | 3 (3) — Grade 1-3 - unlikely to be related
Hemorrhage: nose (Blood and lymphatic system disorders) | 2 (2) — Grade 1-3 - unlikely to be related
Insomnia (General disorders) | 1 (1) — Grade 1-3 - unlikely to be related
International Normalized Ratio of prothrombin time (INR) (Blood and lymphatic system disorders) | 1 (1) — Grade 1-3 - unrelated
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) — Grade 2 - unlikely to be related
Mucositis/stomatitis (Gastrointestinal disorders) | 2 (2) — Grade 1 - unlikely to be related
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) — Grade 1-3 - unrelated
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) — Grade 1-3 - unlikely to be related
Nail changes (Skin and subcutaneous tissue disorders) | 3 (3) — Grade 1-3 - unlikely to be related
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1 (3) — Grade 1-3 - unlikely to be related
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 1 - possibly related
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 1-3 - unrelated
Nausea (Gastrointestinal disorders) | 8 (9) — Grade 1-3 - unlikely to be related
Neuropathy: sensory (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1 - unlikely to be related
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) — Grade 3 - unrelated
Opthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1) — Grade 1-3 - unlikely to be related
Pain - Chest/thorax NOS (General disorders) | 2 (2) — Grade 1-3 - unlikely to be related
Pain - Extremity-limb (General disorders) | 1 (1) — Grade 1 - unlikely to be related
Pain - back (General disorders) | 1 (1) — Grade 1 - unlikely to be related
Pain - head/headache (General disorders) | 1 (1) — Grade 2 - unlikely to be related
Pain - lymph node (General disorders) | 1 (1) — Grade 1 - unrelated
Pain - neck (General disorders) | 1 (1) — Grade 1 - unlikely to be related
Pain - sinus (General disorders) | 1 (1) — Grade 1-3 - unlikely to be related
Pain - stomach (General disorders) | 1 (1) — Grade 1-3 - unlikely to be related
Partial Thromboplastin Time (PTT) (Blood and lymphatic system disorders) | 1 (1) — Grade 1-3 - unrelated
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1 - unrelated
Rigors/chills (General disorders) | 1 (1) — Grade 2 - unrelated
Sodium, serum-low (Metabolism and nutrition disorders) | 1 (1) — Grade 1-3 - unrelated
Sweating (General disorders) | 1 (1) — Grade 1 - unlikely to be related
Taste alteration (Gastrointestinal disorders) | 2 (2) — Grade 1-3 - unlikely to be related
Urine color change (Renal and urinary disorders) | 1 (1) — Grade 1 - unlikely to be related
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1-3 - unlikely to be related
Vomiting (Gastrointestinal disorders) | 4 (6) — Grade 1-3 - unlikely to be related
Weight loss (General disorders) | 1 (1) — Grade 2 - unrelated

LIMITATIONS AND CAVEATS:
This was a Pilot Supportive Care Intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No